CLINICAL TRIAL: NCT03828318
Title: Impact of a Patient-Centered Program for Low Anterior Resection Syndrome a Multicenter Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Collaborators: Providence Healthcare (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Centre Hospitalier du Quebec (Unknown); University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Marylise Boutros, Colorectal Surgeon, Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MP-05-2019-1628
Record Dates: First submitted 2019-01-31; First posted 2019-02-04 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Rectal Cancer; Surgery; Patient Activation; Low Anterior Resection; Low Anterior Resection Syndrome
MeSH Terms: conditions — Rectal Neoplasms; Patient Participation; Low Anterior Resection Syndrome | interventions — Leucine-tRNA Ligase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient Activation Arm (Experimental)
  Interventions: Other: Patient Activation Booklet and nursing support for patients with LARS
- Standard Care Arm (No Intervention)

INTERVENTIONS:
Other: Patient Activation Booklet and nursing support for patients with LARS — The LARS Patient-Centered Program will consist of an educational booklet and nursing support made available only to patients randomized to the intervention group.
  Arms: Patient Activation Arm

SUMMARY:
After undergoing restorative proctectomy for rectal cancer, many patients are left with significant bowel dysfunction, known as Low Anterior Resection Syndrome (LARS). Increased LARS severity correlates with worse perceived global health status and quality of life (QoL). Among patients undergoing rectal resection with a permanent ostomy, there is evidence that supportive and educational interventions improve QoL, ostomy proficiency, self-efficacy and knowledge. However, evidence regarding the impact of such interventions in patients who undergo restorative proctectomy is lacking, despite the latter operation being far more frequently performed.

The overall goal of this study is to evaluate the extent to which a LARS Patient-Centered Program impacts on patient-reported outcome measures (PROMs) after restorative proctectomy for rectal cancer.

This is a randomized-controlled muticenter trial that will include patients who have undergone restorative proctectomy for neoplastic disease (benign or malignant) located in the rectum (0-15cm from the anal verge) with a diverting ostomy and who are scheduled for ostomy closure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>=18 years-old) who have undergone restorative proctectomy for neoplastic disease (benign or malignant) located in the rectum (0-15cm from the anal verge) with a diverting ostomy and who are scheduled for ostomy closure

Exclusion Criteria:

* Patients from whom clear and informed consent cannot be obtained
* Patients unable to read and comprehend English or French
* Patients who cannot be contacted by telephone
* Patients who have undergone major colonic resection in addition to their proctectomy
* Patients on active chemotherapy or radiotherapy treatment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Global quality of life (QoL) | 12 months
  Measured by EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Locations (6):
- Massachusetts General Hospital, Boston, Massachusetts, United States
- Canada (5):
  - Providence Healthcare, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - CHU de Quebec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garfinkle R, Loiselle CG, Park J, Fiore JF Jr, Bordeianou LG, Liberman AS, Morin N, Faria J, Ghitulescu G, Vasilevsky CA, Bhatnagar SR, Boutros M. Development and evaluation of a patient-centred program for low anterior resection syndrome: protocol for a randomized controlled trial. BMJ Open. 2020 May 30;10(5):e035587. doi: 10.1136/bmjopen-2019-035587. PMID 32474427